CLINICAL TRIAL: NCT01664078
Title: A Multicenter, Open Label, Prospective, Non-randomized Study of the InCraft® Stent Graft System in Subjects With Abdominal Aortic Aneurysms (INSPIRATION)
Acronym: INSPIRATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Collaborators: Carelon Research (Other); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P11-4601
Expanded Access: NCT01776450 (No longer available)
Record Dates: First submitted 2012-08-09; First posted 2012-08-14 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2020-08

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- InCraft® - AAA stent graft system (Experimental): Intervention: Endovascular AAA repair using the InCraft device
  Interventions: Device: Endovascular AAA repair with InCraft®

INTERVENTIONS:
Device: Endovascular AAA repair with InCraft®

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of InCraft® in subjects with abdominal aortic aneurysms requiring endovascular repair.

DETAILED DESCRIPTION:
In the US, abdominal aortic aneurysms (AAA) are found in 4-8% of older men and 0.5-1.5% of older women, resulting in 30,000-40,000 elective procedures and 1,400 peri-operative deaths. The most significant complication of AAA is an aneurysm sac rupture from which more than 15,000 patients die annually and is the 15th leading cause of death in elderly between 60 to 85 years of age . In Japan, it is estimated that approximately 14,000 endovascular aneurysm repair (EVAR) and open surgical repair cases were performed in the year 2010 .

Abdominal aortic aneurysms can be treated three ways: (1) Medical management; (2) Open surgical repair; and (3) Endovascular aneurysm repair (EVAR). EVAR has emerged as an alternative treatment of AAA for most patients. It is less invasive than open repair and carries lower rates of early mortality and morbidity . It has also extended treatment options to patients who cannot undergo conventional surgical procedures due to a high operative risk. As EVAR technology evolves, it allows treatment of AAA with increasing complexity of the aortic neck and access vessels.

The InCraft® AAA Stent Graft System is designed for endovascular repair of infrarenal AAAs with complex aortic anatomies. This stent-graft system utilizes nitinol stent and polyester graft technology in an ultra-low profile delivery system, which assists the physician in deploying the device in a controlled, consistent, and precise manner within the aortic neck and iliac arteries. By isolating the aneurysmal sac, the system provides an alternative blood flow path to relieve pressure on the arterial vessel walls and minimize aneurysm growth and the potential for aneurysm sac rupture.

ELIGIBILITY:
Inclusion Criteria:

* Subject must meet ALL of the following inclusion criteria to be enrolled in the study:

  1. Male or Female age 20 years or older;
  2. Proximal aortic neck is 17-31mm in diameter;
  3. Supra-renal aorta, at 20mm above the anticipated landing location, is smaller than the nominal diameter of the aortic bifurcate prosthesis to be used;
  4. Infra-renal aortic neck is ≥10mm in length with supra-renal and infra-renal angulations ≤60°;
  5. Subject has at least one of the following:

     1. AAA size > 5.0 cm;
     2. Increase of the AAA diameter of > 0.5 cm over the last 6 months;
  6. Abdominal treatment length (lowest renal artery origin to the aortic bifurcation) ≥ 9.4cm;
  7. Aortic bifurcation >18mm in diameter;
  8. Iliac landing zone ≥15mm in length;
  9. Iliac landing zone 7-22mm in diameter;
  10. Minimum access vessel size of ≥ 5mm;
  11. Minimum overall AAA treatment length (from lowest renal artery to distal landing zone) of 128 mm;
  12. Women of child bearing potential must be non-pregnant, non-lactating, and not planning to become pregnant during the course of the trial; and have a negative urine or serum pregnancy test within 7 days prior to index procedure;
  13. Provide written informed consent and as applicable written HIPAA authorization (For US sites only) prior to initiation of study procedures;
  14. Willing to comply with the specified follow-up evaluation schedule.

Exclusion Criteria:

* Subjects will be excluded if ANY of the following exclusion criteria apply:

  1. Vascular anatomy in which the placement of the stent-graft will cause occlusion of both internal iliac arteries or necessitates surgical occlusion of both internal iliac arteries;
  2. Subject has one of the following:

     1. Aneurysm sac rupture or leaking abdominal aortic aneurysm;
     2. Mycotic, dissecting, or inflammatory abdominal aortic aneurysm;
     3. Clinically significant acute vascular injury due to trauma;
  3. Significant aortic or iliac mural thrombus, plaque or calcification that would compromise fixation and seal of the device;
  4. A conical aortic neck defined as >3mm distal increase over a 10mm length in the planned seal zone;
  5. Thoracic aortic aneurysm ≥45mm;
  6. Any aortic dissection;
  7. Morbid obesity (BMI >40.0 kg.m2) or other clinical conditions that limit required imaging studies or visualization of the aorta;
  8. Renal insufficiency (Creatinine > 2.0mg/dL) or subject on renal dialysis;
  9. Known allergy or intolerance to nickel titanium (nitinol) , Polyethylene terephthalate (PET), or polytetrafluoroethylene (PTFE);
  10. Known contraindication to undergoing angiography or anticoagulation (e.g. contrast allergies which cannot be treated);
  11. Connective tissue disorder (such as Marfan's Syndrome or Ehlers-Danlos Syndrome);
  12. Coagulopathy, bleeding disorder, or other hypercoagulable state;
  13. Organ transplant recipient or subject requiring systemic immunosuppressant therapy;
  14. Cerebral vascular accident (CVA), MI, or intracranial bleeding within 3 months prior to the procedure;
  15. Active infection or chronic systemic illness at the time of index procedure that may interfere with the study objectives;
  16. Major surgical procedure within 1 month prior to the index procedure or pre-planned within 1 month afterwards;
  17. Co-existing condition with a life expectancy of less than 2 years at time of procedure;
  18. Current or planned participation in any other investigational drug or medical device clinical study that has not completed primary endpoint(s) evaluation;
  19. Existing AAA surgical graft and/or a AAA stent-graft system;
  20. Other medical, social, or psychological issues that in the opinion of the investigator preclude the subjects from receiving this treatment, and the procedures and evaluations pre- and posttreatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2018-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel S Makaroun, MD, Principal Investigator — University of Pittsburgh; Takao Ohki, MD, Principal Investigator — Jikei University School of Medicine
Locations (2):
- Michel S. Makaroun, MD, Pittsburgh, Pennsylvania, United States
- Takao Ohki, MD, Minato-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iantorno M, Buchanan KD, Bernardo NL, Torguson R, Waksman R. Overview of the 2018 US Food and Drug Administration Circulatory System Devices Panel meeting on the INCRAFT AAA Stent Graft System. Cardiovasc Revasc Med. 2019 May;20(5):403-408. doi: 10.1016/j.carrev.2019.02.018. Epub 2019 Feb 18. PMID 30879790

RESULTS

PARTICIPANT FLOW:
Groups:
- InCraft® - AAA Stent Graft System: Intervention: Endovascular AAA repair using the InCraft device
  Endovascular AAA repair with InCraft®
Period: Overall Study
Arm/Group | InCraft® - AAA Stent Graft System
Started | 190
Completed | 121
Not Completed | 69
Not completed — Death | 9
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 2
Not completed — missed 5 year visit | 1
Not completed — Other | 53

BASELINE CHARACTERISTICS:
Arm/Group | InCraft® - AAA Stent Graft System
Number analyzed (Participants) | 190
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Analysis was split between male and female measurements.
  years
    Male: number analyzed (Participants) | 171
    Male | 73.6 (7.58)
    Female: number analyzed (Participants) | 19
    Female | 75.3 (7.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 171
Region of Enrollment [Number; unit: participants]
  United States | 134
  Japan | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of MAE (Major Adverse Events) Based Upon a Composite MAE Rate
Description: defined as a composite of:
  * Death
  * Stroke
  * Myocardial Infarction
  * New Onset Renal Failure (requiring dialysis)
  * Respiratory Failure (requires mechanical ventilation)
  * Paralysis/paraparesis
  * Bowel ischemia (requiring surgical intervention)
  * Procedural blood loss ≥1,000 cc
Time Frame: 30 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | InCraft® - AAA Stent Graft System
Number analyzed (Participants) | 183
Participants | 20
Statistical Analysis 1: Comparison: InCraft® - AAA Stent Graft System; Test type: Other — The Intent-to-Treat (ITT) analysis set includes all subjects who had the aortic bifurcate device introduced into the body. This ITT analysis set will be used for all safety and clinical assessment endpoints; p = 0.47, Mixed Models Analysis

2. Primary Outcome: Number of Participants With Successful Aneurysm Treatment
Description: Successful aneurysm treatment which is a composite endpoint of the following:
  * Technical Success at the conclusion of the index procedure, defined as successful insertion of the delivery system through the vasculature and successful deployment of the device at the intended location. The endovascular graft must be patent, with absence of types I or III endoleaks or aneurysm sac rupture, at the time of procedure completion as confirmed by angiography or other imaging modality;
  * Absence of post-operative aneurysm enlargement (growth > 5 mm) or stent graft migration (> 10mm) compared to the one month size measurement at anytime up to 1-year;
  * Absence of post-operative conversion to open surgery, sac rupture, endoleak Type I / III, or graft occlusion (including unilateral or bilateral limb occlusion) at any time up to 1-year.
Time Frame: Up to 1 year post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | InCraft® - AAA Stent Graft System
Number analyzed (Participants) | 173
Participants | 152

3. Secondary Outcome: Procedure-related Complications
Description: Adverse events that are a result of the procedure itself.
Time Frame: Through 1 month, 180-days, 360-days and annually to 5-years post-procedure
Measure: Count of Participants; unit: Participants
Groups:
- Site-reported Procedure-related AEs Through 1 Month; Site-reported Procedure-related AEs Through 180 Days; Site-reported Procedure-related AEs Through 360 Days; Site-reported Procedure-related AEs Through 2 Years; Site-reported Procedure-related AEs Through 3 Years; Site-reported Procedure-related AEs Through 4 Years; Site-reported Procedure-related AEs Through 5 Years: procedure-related complications were tabulated as secondary safety endpoints
Arm/Group | Site-reported Procedure-related AEs Through 1 Month | Site-reported Procedure-related AEs Through 180 Days | Site-reported Procedure-related AEs Through 360 Days | Site-reported Procedure-related AEs Through 2 Years | Site-reported Procedure-related AEs Through 3 Years | Site-reported Procedure-related AEs Through 4 Years | Site-reported Procedure-related AEs Through 5 Years
Number analyzed (Participants) | 190 | 189 | 188 | 186 | 185 | 185 | 186
Participants | 98 | 100 | 104 | 104 | 109 | 112 | 113

4. Secondary Outcome: Aneurysm-related Mortality
Time Frame: At 30-days, 180-days, 360-days and annually to 5-years post-procedure
Measure: Count of Participants; unit: Participants
Groups:
- Aneurysm-related Morality Through 1 Month; Aneurysm-related Morality Through 180 Days; Aneurysm-related Morality Through 360 Days; Aneurysm-related Morality Through 2 Years; Aneurysm-related Morality Through 3 Years; Aneurysm-related Morality Through 4 Years; Aneurysm-related Morality Through 5 Years: Aneurysm-related mortality is defined as death from AAA rupture, or death within 30 days of open aortic surgical or endovascular repair, or death from any subsequent procedure required to treat the same aneurysm.
Arm/Group | Aneurysm-related Morality Through 1 Month | Aneurysm-related Morality Through 180 Days | Aneurysm-related Morality Through 360 Days | Aneurysm-related Morality Through 2 Years | Aneurysm-related Morality Through 3 Years | Aneurysm-related Morality Through 4 Years | Aneurysm-related Morality Through 5 Years
Number analyzed (Participants) | 190 | 187 | 183 | 176 | 172 | 168 | 165
Participants | 1 | 1 | 1 | 1 | 1 | 1 | 1

5. Secondary Outcome: Incidence of Secondary Interventions
Description: The incidence of secondary interventions within 1 year post-procedure, needed to prevent the occurrence of a significant event. Significant event being defined as: aneurysm enlargement (growth > 5 mm), stent graft migration (> 10mm) compared to the one month size, endoleak type I / III, graft occlusion, sac rupture.
Time Frame: through 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Secondary Intervention Through 1 Month; Secondary Intervention Through 180 Days; Secondary Intervention Through 360 Days; Secondary Intervention Through 2 Years; Secondary Intervention Through 3 Years; Secondary Intervention Through 4 Years; Secondary Intervention Through 5 Years: The incidence of secondary interventions within 1 year post-procedure, needed to prevent the occurrence of a significant event. Significant event being defined as: aneurysm enlargement (growth > 5 mm), stent graft migration (> 10mm) compared to the one month size, endoleak type I / III, graft occlusion, sac rupture.
Arm/Group | Secondary Intervention Through 1 Month | Secondary Intervention Through 180 Days | Secondary Intervention Through 360 Days | Secondary Intervention Through 2 Years | Secondary Intervention Through 3 Years | Secondary Intervention Through 4 Years | Secondary Intervention Through 5 Years
Number analyzed (Participants) | 189 | 183 | 176 | 162 | 149 | 132 | 118
Participants | 1 | 5 | 8 | 7 | 12 | 8 | 4

6. Secondary Outcome: Major Adverse Events (MAEs) and Individual Components of the MAEs
Time Frame: At 180-days, 360-days and annually to 5-years post-procedure
Measure: Count of Participants; unit: Participants
Groups:
- MAEs Through 180 Days; MAEs Through 360 Days; MAEs Through 2 Years; MAEs Through 3 Years; MAEs Through 4 Years; MAEs Through 5 Years: All MAEs are site-reported then adjudicated by the CEC.
Arm/Group | MAEs Through 180 Days | MAEs Through 360 Days | MAEs Through 2 Years | MAEs Through 3 Years | MAEs Through 4 Years | MAEs Through 5 Years
Number analyzed (Participants) | 187 | 183 | 176 | 172 | 168 | 165
Participants
  Death | 3 | 6 | 12 | 22 | 35 | 45
  Stroke | 3 | 4 | 9 | 13 | 15 | 17
  Myocardial infarction | 3 | 6 | 7 | 9 | 12 | 13
  New onset renal failure (requiring dialysis) | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory failure (requiring mechanical ventilat | 1 | 2 | 2 | 2 | 2 | 2
  Paralysis / paraparesis | 0 | 0 | 0 | 0 | 0 | 0
  Bowel ischemia (requiring surgical intervention) | 0 | 0 | 0 | 0 | 0 | 1
  Procedural blood loss (≥1,000 cc) | 4 | 4 | 4 | 4 | 4 | 4

7. Secondary Outcome: Device-related Events
Description: Endoleak(s), Aneurysm sac rupture, Fracture(s, Delivery System Malfunction, Device Malfunction, Stent Graft Migration - evidence of proximal or distal movement of the stent graft >10mm relative to fixed anatomic landmarks compared with 1 month, Graft Occlusion (including unilateral or bilateral limb occlusion, Conversion to open surgery, and Aneurysm Enlargement - defined as an increase in maximum aneurysm cross sectional diameter > 5mm compared to the 1-month measurement.
Time Frame: At 1 month, 6 months, 1 year and annually to 5-years post-procedure
Measure: Count of Participants; unit: Participants
Groups:
- Device-related Events Through 1 Month; Device-related Events Through 180 Days; Device-related Events Through 360 Days; Device-related Events Through 2 Years; Device-related Events Through 3 Years; Device-related Events Through 4 Years; Device-related Events Through 5 Years: Endoleak(s), Aneurysm sac rupture, Fracture(s, Delivery System Malfunction, Device Malfunction, Stent Graft Migration - evidence of proximal or distal movement of the stent graft >10mm relative to fixed anatomic landmarks compared with 1 month, Graft Occlusion (including unilateral or bilateral limb occlusion, Conversion to open surgery, and Aneurysm Enlargement - defined as an increase in maximum aneurysm cross sectional diameter > 5mm compared to the 1-month measurement.
Arm/Group | Device-related Events Through 1 Month | Device-related Events Through 180 Days | Device-related Events Through 360 Days | Device-related Events Through 2 Years | Device-related Events Through 3 Years | Device-related Events Through 4 Years | Device-related Events Through 5 Years
Number analyzed (Participants) | 181 | 167 | 159 | 141 | 131 | 115 | 104
Participants | 0 | 7 | 16 | 24 | 40 | 42 | 48

8. Secondary Outcome: Technical Success Confirmed by CT or Other Imaging Modality
Description: The study evaluated technical success at 30-days as one of the secondary effectiveness endpoints. The definition of technical success is defined as patency of the endovascular graft, with the absence of Type I or III endoleaks or aneurysm sac rupture, up to 30-days post-procedure completion as confirmed by CT or other imaging modality.
Time Frame: At 30-days
Measure: Count of Participants; unit: Participants
Groups:
- Technical Success: Technical success confirmed by CT or other imaging modality
Arm/Group | Technical Success
Number analyzed (Participants) | 188
Participants | 188

9. Secondary Outcome: Length of Hospital Stay (Days) Post Index Procedure
Time Frame: up to 17 days
Measure: Mean (Standard Deviation); unit: days
Groups:
- Length of Hospital Stay (Days) Post Index Procedure: Length of hospital stay (days) post index procedure as part of the clinical utility measure
Arm/Group | Length of Hospital Stay (Days) Post Index Procedure
Number analyzed (Participants) | 190
days | 2.7 (2.88)

10. Secondary Outcome: Length of Intensive Care Unit (ICU) Stay (Hours) Post Index Procedure
Time Frame: up to 48 hours
Measure: Mean (95% Confidence Interval); unit: hours
Groups:
- Length of Intensive Care Unit (ICU) Stay (Hours) Post Index pr: Length of Intensive Care Unit (ICU) stay (hours) post index pr as part of the clinical utility measure
Arm/Group | Length of Intensive Care Unit (ICU) Stay (Hours) Post Index pr
Number analyzed (Participants) | 190
hours | 8 [0 to 18.59]

11. Secondary Outcome: Length of the Index Procedure (Minutes)
Time Frame: 1 day
Measure: Mean (95% Confidence Interval); unit: minutes
Groups:
- Length of the Index Procedure (Minutes): Length of the Index Procedure (Minutes) as part of the clinical utility measure
Arm/Group | Length of the Index Procedure (Minutes)
Number analyzed (Participants) | 190
minutes | 102.7 [58.83 to 146.57]

12. Other Pre Specified Outcome: Pain Post-Operatively
Description: Outcome measured by the SF36v2 Health Status Survey where all items are scored so that a high score defines a more favorable health state. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Time Frame: Baseline, 1 month, 6 months and 1 year post-procedure
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Groups:
- Pain Post-Operatively at Baseline: Pain post-operatively as measured by the SF36v2 (bodily pain BP) at screening, 1-month, 6-months, and 1-year follow-up
- Pain Post-Operatively at 1-Month; Pain Post-Operatively at 6-Months; Pain Post-Operatively at 1-Year: Pain post-operatively were compared to baseline values, as measured by the SF36v2 (bodily pain BP) at screening, 1-month, 6-months, and 1-year follow-up
Arm/Group | Pain Post-Operatively at Baseline | Pain Post-Operatively at 1-Month | Pain Post-Operatively at 6-Months | Pain Post-Operatively at 1-Year
Number analyzed (Participants) | 187 | 188 | 179 | 175
Units on a Scale | 71.4 [45.18 to 97.62] | 70.2 [44.7 to 95.7] | 71.5 [43.9 to 99.1] | 73.1 [47.68 to 98.52]

13. Other Pre Specified Outcome: Physical Functioning Post-operatively
Description: Physical Functioning (PF) Outcome measured by the SF36v2 Health Status Survey where all items are scored so that a high score defines a more favorable health state. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Time Frame: Screening, 1 month, 6 months and 1 year post-procedure
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Groups:
- Physical Functioning Post-operatively at Baseline; Physical Functioning Post-operatively at 1 Month; Physical Functioning Post-operatively at 6 Month; Physical Functioning Post-operatively at 1 Year: Physical functioning post-operatively as measured by the SF36v2 [physical component summary (PCS), physical functioning (PF) and role physical (RP) domains] at screening, 1-month, 6-months, and 1-year follow up
Arm/Group | Physical Functioning Post-operatively at Baseline | Physical Functioning Post-operatively at 1 Month | Physical Functioning Post-operatively at 6 Month | Physical Functioning Post-operatively at 1 Year
Number analyzed (Participants) | 188 | 188 | 179 | 175
Units on a Scale | 69.2 [42.96 to 95.44] | 66.5 [38.93 to 94.07] | 68.6 [41.43 to 95.77] | 68.2 [41.49 to 94.91]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from index procedure until completion of study or early termination.
Description: All-Cause Mortality, Serious Adverse Events, Other (Not Including Serious) Adverse Events.
Groups:
- InCraft: Infrarenal Abdominal Aortic Aneurysm Stent Graft System
Arm/Group | InCraft
All-Cause Mortality (participants affected / at risk) | 45/188
Serious Adverse Events (participants affected / at risk) | 52/188
Other Adverse Events (participants affected / at risk) | 93/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | InCraft (N=188)
Cardiac disorders (Cardiac disorders) | 15
Congenital disorders (Congenital, familial and genetic disorders) | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 5
General disorders and administration site conditions (General disorders) | 7
Infections and infestations (Infections and infestations) | 2
Injury, poisoning and procedural complications2 (Injury, poisoning and procedural complications) | 6
Investigations (Investigations) | 1
Neoplasms benign, malignant and unspecified (including cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Nervous system disorders (Nervous system disorders) | 9
Renal and urinary disorders (Renal and urinary disorders) | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 6
Vascular disorders (Vascular disorders) | 9
Blood and Lymphatic (Blood and lymphatic system disorders) | 2
Metabolisms and Nutrition Disorders (Metabolism and nutrition disorders) | 3
Surgical and medical procedures (Surgical and medical procedures) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | InCraft (N=188)
Gastrointestinal disorders (Gastrointestinal disorders) | 15
General disorders and administration site conditions (General disorders) | 15
Infections and infestations (Infections and infestations) | 10
Injury, poisoning and procedural complications1 (Injury, poisoning and procedural complications) | 15
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 14
Nervous system disorders (Nervous system disorders) | 11
Renal and urinary disorders (Renal and urinary disorders) | 13
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 16
Vascular disorders4 (Vascular disorders) | 20

LIMITATIONS AND CAVEATS:
Number of participants at risk my vary depending on varying windows used for analysis, imaging availability, visits completed and will therefore not be consistent throughout report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No